CLINICAL TRIAL: NCT06575153
Title: A Phase 1, Randomized, Double-blind, Single Ascending Dose and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ART5803 Compared With Placebo in Healthy Participants
Brief Title: Phase 1 Study of ART5803 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arialys Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ART5803-101
Record Dates: First submitted 2024-08-15; First posted 2024-08-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autoimmune Encephalitis
Keywords: Anti-N-methyl-D-aspartate receptor (NMDAR); Encephalitis; Anti-N-methyl-D-aspartate receptor (NMDAR) Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Encephalitis

STUDY DESIGN:
Intervention Model Description: This study will include up to 5 cohorts in Part 1 (SAD) and up to 3 cohorts in Part 2 (MAD). Each cohort will consist of 8 participants who will receive a single IV dose of either ART5803 or placebo (6 active [ART5803], 2 placebo) based on the individual participant's randomly assigned treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 (SAD) Cohort 1 - Dose Level 1 (Experimental): 3 mg/kg of ART5803 IV infusion over approximately 90 minutes (±60 minutes)
  Interventions: Drug: ART5803
- Part 1 (SAD) Cohort 2- Dose Level 2 (Experimental): 10 mg/kg of ART5803 IV infusion over approximately 90 minutes (±60 minutes)
  Interventions: Drug: ART5803
- Cohort 3 (SAD)/Cohort A (MAD) - Dose Level 3 (Experimental): 30 mg/kg of ART5803 IV infusion over approximately 90 minutes (±60 minutes)
  Interventions: Drug: ART5803
- Cohort 4 (SAD)/Cohort B (MAD) - Dose Level 4 (Experimental): 60 mg/kg of ART5803 IV infusion over approximately 90 minutes (±60 minutes)v
  Interventions: Drug: ART5803
- Cohort 5 (SAD)/Cohort C (MAD) - Dose Level 5 (Experimental): 100 mg/kg of ART5803 IV infusion over approximately 90 minutes (±60 minutes)
  Interventions: Drug: ART5803
- Placebo (No Intervention): 0.9% normal saline IV infusion over approximately 90 minutes (±60 minutes)

INTERVENTIONS:
Drug: ART5803 — A monovalent (one-armed) antibody, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor.
  Arms: Cohort 3 (SAD)/Cohort A (MAD) - Dose Level 3; Cohort 4 (SAD)/Cohort B (MAD) - Dose Level 4; Cohort 5 (SAD)/Cohort C (MAD) - Dose Level 5; Part 1 (SAD) Cohort 1 - Dose Level 1; Part 1 (SAD) Cohort 2- Dose Level 2

SUMMARY:
The study is a Phase 1, single-center, randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, pharmacokinetics (PK), and immunogenicity of ART5803 compared with placebo in healthy adult participants

DETAILED DESCRIPTION:
Anti-N-methyl-D-aspartate receptor (NMDAR) encephalitis is one of the most common causes of autoimmune encephalitis. The disease is caused by the development of autoantibodies against the amino (N)-terminal domain (NTD) of the NMDAR subunit 1 (NR1) that bind and cross link the receptors, leading to receptor internalization and loss of function. Arialys has developed a monovalent (one-armed) antibody, ART5803, that binds to the NTD of the NMDAR NR1 subunit without causing NMDAR inhibition, activation, or receptor internalization, while simultaneously blocking the ability of the pathogenic anti-NMDAR autoantibodies to bind to the receptor. This first-in-human (FIH) study will assess the safety, tolerability, pharmacokinetics (PK), and immunogenicity of ART5803 compared with placebo in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a male or female, 18 to 65 years of age, inclusive, at the time of informed consent and has a body mass index (BMI) of ≥18 to ≤32 kg/m²
2. The participant is healthy, as determined by medical history, physical examinations, and the clinical Investigator's judgment.
3. The participant must be willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
4. The participant must be willing and able to comply with all study procedures.
5. Sexually active female participants of childbearing potential and male participants with female partner(s) of childbearing potential must be willing to use a highly effective method of contraception while participating in the study.
6. Female participants of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who are surgically sterile (surgical bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) confirmed by medical history or are post-menopausal (i.e., no menstrual bleeding for more than 12 months without an alternative medical cause and confirmation with more than 1 follicle-stimulating hormone measurement of at least > 40 IU/L [or higher per local institutional guidelines]).Women of non-childbearing potential are not required to use any contraceptive method.
7. Male participants with female partners of childbearing potential must agree to use highly effective methods of contraception, from study drug administration until at least 90 days after the last study drug administration.
8. Male participants must agree not to donate sperm and female participants must agree not to donate eggs, for the duration of the study and until at least 90 days after the last study drug administration.
9. Participants must agree to not donate blood for at least 3 months after the end-of-study (EOS) visit

Exclusion Criteria:

1. The participant is pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
2. The participant has used an investigational product or investigational medical device within 30 days prior to Screening, or is required to use any investigational agent prior to completion of all scheduled study assessments.
3. Has a condition of such severity and acuity, in the opinion of the Investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study.
4. The participant has a history of cancer, apart from squamous cell carcinoma of the skin or basal cell carcinoma of the skin. Squamous cell and basal cell carcinomas should be treated with documented success of curative therapy >3 months prior to randomization.
5. The participant has any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality, which may interfere with the evaluation or administration of the study drug, interpretation of participant safety or study results, or would make participation in the study an unacceptable risk including any significant acute or chronic medical condition. It is the responsibility of the Investigator to assess the clinical significance; however, consultation with the medical monitor may be warranted.
6. Has a concurrent disease or condition that, in the view of the Principal Investigator, places the participant at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety. Participants with fully resolved childhood asthma that has had no reoccurrences or hospitalizations remain eligible for participation.
7. The participant is a regular smoker (cigarettes, e-cigarettes, and vaping included), defined as smoking daily. Participants that are non-daily smokers (up to ≤5 cigarettes per week [or vaping or e-cigarette equivalent]) are permitted to participate in the study and must agree to refrain from smoking from 2 weeks before the first study drug administration until the end of the inpatient stay (Part 1: Day 5; Part 2: Day 29).
8. The participant has a contraindication to undergo LP, including international normalized ratio (INR) >1.4 or other coagulopathy, platelet cell count of <120,000/µL, infection at the desired LP site, current use of anti-coagulant medication except for low dose acetylsalicylic acid, degenerative arthritis, spinal scoliosis, back surgery, suspected increased intracranial pressure on history or neurologic exam, non-communicating hydrocephalus or intracranial mass, or prior history of spinal mass or trauma.
9. The participant has severe drug allergic history or anaphylaxis to 2 or more food products or medicines (including known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine, methylprednisolone or equivalent glucocorticoid, or lidocaine).
10. The participant has a known history of allergy or reaction to any component of the investigational agent formulation or placebo, or history of anaphylaxis following any biologic therapy.
11. The participant has a history of alcohol abuse or drug addiction in the past 12 months.
12. The participant has undergone significant trauma or major surgery within 4 weeks of Screening.
13. The participant has had a vaccination with live virus, attenuated live virus, or any live viral components within 2 weeks prior to study drug administration or is planning to receive these vaccines at any time during the study and up to 8 weeks following the last study drug administration.
14. The participant has ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

    1. Serum creatinine level more than 1.25× upper limit of normal (ULN) or an estimated glomerular filtration rate value <80 mL/min/1.73 m² calculated with the Chronic Kidney Disease Epidemiology Collaboration formula and more than trace protein in urine.
    2. Total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values more than >2×ULN. Note: participants with a history of Gilbert's syndrome are excluded from participation in the study.
    3. Hematological or coagulation values outside the normal reference range for local laboratory results unless regarded as clinically not significant.
    4. Confirmed positive test for hepatitis B serology (hepatitis B surface antigen and core antibody) and/or hepatitis C polymerase chain reaction.
15. The participant has a 12-lead ECG demonstrating corrected QT interval by Fridericia (QTcF) >450 ms. If QTcF exceeds 450 ms the ECG should be repeated 2 more times and the average of the 3 QTcF values should be used to determine the participant's eligibility.
16. The participant has Investigator determined coronavirus disease of 2019 (COVID-19) within 4 weeks prior to Day -1, received the COVID-19 vaccine within 2 weeks prior to study drug administration, or plans to receive a COVID-19 vaccine within 9 weeks after study drug administration. Regional and site COVID-19 testing policies should be followed throughout the study.
17. The participant has a positive urine or blood result for drugs of abuse (defined as any illicit drug use) at Screening or check-in (Day -1).
18. The participant has received any NMDAR modulator other than the study drug (e.g., ketamine, memantine, dextromethorphan, amantadine, ifenprodil, phencyclidine [PCP], acamprosate, D-cycloserine) or IVIG from within 30 days or 5 half-lives of the other NMDAR modulator or IVIG (whichever is longer) of study drug administration until the end of the study.
19. The participant has a known history of a primary immunodeficiency (congenital or acquired) or an underlying condition such as human immunodeficiency virus infection
20. The participant has had a bacillus of Calmette and Guérin vaccine within 1 year of enrollment.
21. The participant has a history of severe depression, bipolar disease, or schizophrenia.
22. The participant has a risk of suicide per the C-SSRS (a score of 4 or 5 on ideation or any suicidal behavior) or according to the Investigator's clinical judgment, has made a suicide attempt in the previous 6 months, or has a history of deliberate self-harm in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Safety will be assessed by the incidence and severity of treatment-emergent adverse events (TEAEs) | 12 weeks
  ART5803 safety, as measured by the number of treatment emergent adverse events compared with placebo.
Safety will be assessed by clinically significant changes in physical and neurological examination findings | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes in physical and neurological examination findings compared with placebo.
Safety by assessed by clinically significant changes in vital signs | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes in vital signs including systolic and diastolic blood pressure, pulse rate, respiration rate, and body temperature as compared to placebo.
Safety by assessed by clinically significant changes in clinical laboratory outcomes | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes in clinical laboratory outcomes including clinical chemistry, hematology, coagulation, and urinalysis as compared to placebo.
Safety by assessed by clinically significant changes in 12-lead ECG findings | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes 12-lead ECG findings as compared to placebo.
Safety by assessed by clinically significant changes in concomitant medications | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes in concomitant medications as compared to placebo.
Safety by assessed by clinically significant changes in presence of anti-drug antibodies (ADAs) | 12 weeks
  ART5803 safety, will be assessed by clinically significant changes in presence of anti-drug antibodies (ADAs) as compared to placebo.
Safety will be assessed by incidence of dose-limiting toxicity (DLTs) | 12 weeks
  ART5803 safety, will be assessed by incidence of dose-limiting toxicity (DLTs) as compared to placebo.
Safety will be assessed by change in suicidal tendency measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | 12 weeks
  ART5803 safety, will be assessed by change in suicidal tendency as measured by the incidence of positive responses (Yes) to Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) as compared to placebo.

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by maximum concentration (Cmax) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by minimum concentration (Cmin) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by time at which Cmax is observed (tmax) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by area under the curve from time 0 to the last measurable concentration (AUC0-t) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by area under the curve from time 0 extrapolated to infinity (AUC0-∞) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by the half-life (t½) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by the volume of distribution (Vd) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To characterize and compare the PK profile of single ascending IV doses and multiple ascending IV doses of ART5803 as measured by clearance (CL) as compared with placebo.
To assess the pharmacokinetics (PK) of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Serum collected over 96 hours after administration, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, and Day 85; CSF collected 48 hours after administration, Day 29 and Day 43
  To asses the CSF/serum ratio of ART5803 at multiple time points.

OTHER OUTCOMES:
To assess changes in cognition as measured by the Mini-Mental State Examination (MMSE) after single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Day 1 (pre-dose), 24 hours after administration, Day 8, Day 29, Day 57, and Day 85
  To assess the change in MMSE total scores from baseline as compared with placebo.
To assess changes in cognition as measured by the Trial Making Test Part A & B (TMT-A and TMT-B) after single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Day 1 (pre-dose), 24 hours after administration, Day 8, Day 29, Day 57, and Day 85
  To assess the change in TMT-A and TMT-B total scores from baseline as compared with placebo.
To assess the immunogenicity of single ascending IV doses and multiple ascending IV doses of ART5803 compared with placebo | Day 1 (pre-dose), Day 8, Day 29, Day 43, Day 71, and Day 85
  To assess the incidence of anti-drug antibodies (ADAs) in serum from single ascending IV doses and multiple ascending IV doses of ART5803 as compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sankalp Gokhale, MD, MBA, Study Chair — Arialys Therapeutics
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No